CLINICAL TRIAL: NCT06798233
Title: Development and Validation of a New Questionnaire for Caregivers to Assess Hip Pain in Quadriplegic Pediatric Patients: Non-Ambulatory Hip Pain Questionnaire
Acronym: NAHPq
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: IRCCS Fondazione Stella Maris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 254/2024/SPER/AUSLRE
Record Dates: First submitted 2025-01-03; First posted 2025-01-29 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-01

CONDITIONS: Quadriplegia/Tetraplegia
Keywords: hip pain; pain measurements; children; adolescents; cerebral palsy
MeSH Terms: conditions — Quadriplegia; Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The study includes the following steps:
  * development of the questionnaire to identify hip pain by means of a Delphi Method approach, involving a group of experts (clinicians and caregivers)
  * validation of the questionnaire by administering it to 100 caregivers of quadriplegic non-communicative patients
  * comparing results of the questionnaire with r-FLACC scale filled out by the physiatrist moving the hip during the visit
Masking Description: * Participants are the caregivers that will fill out the questionnaire aimed at "diagnosing" their child's hip pain: they cannot be masked.
  * The physiatrist will verify the presence of hip pain while moving the hip during the visit, and assess it by means of the r-FLACC scale: he/she will be masked to the questionnaire.
  * The statistician will examine pooled data and compare the questionnaires with r-FLACC scale: he/she will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with quadriplegia (Experimental): Care givers of patients with quadriplegia will fill out a questionnaire aimed at identifying hip pain
  Interventions: Diagnostic Test: Non-Ambulatory Hip Pain questionnaire

INTERVENTIONS:
Diagnostic Test: Non-Ambulatory Hip Pain questionnaire — a new questionnaire for care givers to identify hip pain in pediatric patients with quadriplegia

SUMMARY:
The goal of this clinical trial is twofold:

1. to develop a questionnaire for care givers to assess hip pain in quadriplegic pediatric patients who are not able to communicate it independently
2. to validate this questionnaire in a cohort of 100 pediatric patients with quadriplegia

Researchers will :

1. involve 10 experts (8 multiprofessional clinicians and 2 parents) in a Delphi approach to develop the questionnaire
2. assess construct validity and reliability of the questionnaire submitting it to 100 care givers of pediatric patients with quadriplegia, and comparing results with the Revised Face Legs Activity Cry and Consolability (r-FLACC) Scale assessed by the physiatrist during the visit

Participants will:

1. as experts, firstly answer open questions on this topic, secondly evaluate each item of the new questionnaire by means of a 5-point Liekert scale
2. as caregivers of pediatric patients with quadriplegia, fill out the questionnaire within 2 weeks after the visit

DETAILED DESCRIPTION:
Patients with quadriplegia have complex health and care needs: multimorbidity increases mortality, worsens functioning and participation (according to the ICF model) and negatively affects quality of life. One of the main problems that is difficult to identify early is undoubtedly pain, complicated by the many potential sources of pain and the different levels of intellectual and communicative disability of these patients. Although pain is a frequent concern for these patients and their families, as it greatly interferes with the daily activities and quality of life of all members of the household, it is very often underestimated, consequently little treated and little studied. In the pediatric population, the majority of patients with these characteristics have a diagnosis of Cerebral Palsy (CP): 26% have quadriplegia, classifiable as level IV-V of the Gross Motor Function Classification System (GMFCS). In children with CP, pain is a secondary problem to primary disorders, but with a strongly negative impact on the overall picture, both for the strictly clinical aspects and for the deterioration of quality of life. More than 90% of children with CP between 5 and 18 years of age report experiences of pain within the 1st year (48% ambulatory patients, 79% non-ambulatory patients). A previous study on a sample of 101 parents of children with nonverbal CP, between 2 and 20 years old, report that 65% reported painful experiences in the last 4 weeks (for 17% the pain is intense, for 28% it is daily). Among the most common causes of chronic pain is described pain of musculoskeletal origin, often caused by joint misalignments, increased muscle tone and osteoporosis. Hip dislocation and associated pain are certainly among the main topics of rehabilitation relevance. According to literature data, the specific prevalence of hip pain ranges from 9.6% to 27% in non-ambulatory children or adolescents with CP. Hip pain increases with age, GMFCS level, and degree of dislocation. To monitor and detect hip migration early, as well as to prevent pain, several countries have developed specific hip surveillance programs for children with CP. Population-based registry studies have reported a prevalence of hip pain of 7.9% in patients with IV GMFCS and 20.5% among patients with IV GMFCS in the 4-16 age group, and an overall prevalence of 72% among adolescents and young adults with PC. The highest prevalence of hip pain is found in patients over 11 years of age. In non-verbal children or children with limited verbal and cognitive abilities, the description of pain is entrusted to parents and/or caregivers (observational/proxy methods), who know and interpret the typical behavioral response of their child. Therefore, in addition to a detailed medical history and physical examination, the importance of recognizing painful behaviors and the use of pain hetero-assessment scales was highlighted. According to a recent systematic review the parent or caregiver report can be used as an alternative for pain assessment in children with or at high risk of CP. The NICE guidelines for the identification of pain and the assessment of its intensity in children and adolescents with communication difficulties suggest the use of the Paediatric Pain Profile (PPP) or the Non-communicating Children's Pain Checklist - postoperative version (NCCPC-R). However, none of these tools are specific to CP patients. In 2004 the Pain Assessment Instrument for Cerebral Palsy (PAICP) was presented, a questionnaire dedicated to patients with severe CP, which uses Alternative Augmentative Communication images to identify potentially painful situations associated with the Faces Pain Scale to identify pain intensity. This tool, however, is not specific for hip pain and, moreover, implies a sufficient cognitive level to use the aforementioned communication tools. Based on our knowledge, there are no new studies that point to specific and/or effective tools for the identification of hip pain in quadriplegic pediatric patients. Therefore, to date, there is no specific assessment tool available for this population that investigates the presence and characteristics of hip pain. The aim of the present study is to develop and validate a questionnaire to be administered to caregivers, that can assist healthcare professionals in the identification of hip pain in pediatric patients with quadriplegia.

ELIGIBILITY:
Inclusion Criteria:

* GMFCS IV-V
* CFCS III-V
* subscription of consent

Exclusion Criteria:

* care givers not speaking Italian or English

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Content validity of the Non-Ambulatory Hip Pain questionnaire (NAHPq) | The NAHPq is filled out by the caregiver within 2 weeks after the recruitment visit, during which the hip pain is assessed by the physiatrist with the r-FLACC scale.
  The questionnaire developed by means of the Delphi Method will be submitted to a group of 8-10 experts. They will evaluate each item and attribute one of the following judgments "essential", "usefull but not essential" or "unnecessary". The content validity ratio (CVR) for each item and the overall content validity index (CVI) will be calculated. The CVI is expected to be > 0.75 for eight-expert group or > 0.62 for 10-expert group. In case of lower values the items with the lowest CVR values will require to be revised, considering the experts' comments. The minimum and maximum values of the NAHPq are to be defined during the development Delphi phase; higher values will represent higher pain.
Internal reliability of the Non-Ambulatory Hip Pain questionnaire (NAHPq) | The NAHPq is filled out by the caregiver within 2 weeks after the recruitment visit, during which the hip pain is assessed by the physiatrist with the r-FLACC scale.
  After validity assessment, the questionnaire will be submitted to 100 caregivers of quadriplegic non-communicative patients aged 1-20 years. The Pearson's coefficient will be used to assess the inter-item correlation and the item-to-total correlation. The Cronbach's alpha will be calculated to measure the internal consistency.

SECONDARY OUTCOMES:
Criterion validity of the Non-Ambulatory Hip Pain questionnaire (NAHPq) | The hip pain will be assessed by the physiatrist with the r-FLACC scale during the visit; by the care giver with the NAHPq within 2 weeks after the visit.
  Measure of the degree of reproducibility of the pain assessment with the questionnaire completed by the families compared to the clinical assessment of pain performed by the clinician during the visit by means of the Revised Face Legs Activity Cry and Consolability (r-FLACC) Scale (minimum value 0, maximum value 10; higher scores mean a worse outcome). The agreement between the NAHPq and the FLACC scale will be measured by means of Cohen's kappa coefficient or another correlation coefficient.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Fondazione Stella Maris, Pisa, Italy
  - AziendaUSL IRCCS Reggio Emilia, Spilamberto, Modena

IPD SHARING:
Plan to Share IPD: No
The IPD after conclusion of this study will be made available by the authors upon reasonable request.The data are not publicly available due to restrictions (e.g., their containing information that could compromise the privacy of research participants)

REFERENCES:
- [Background] Hidecker MJ, Paneth N, Rosenbaum PL, Kent RD, Lillie J, Eulenberg JB, Chester K Jr, Johnson B, Michalsen L, Evatt M, Taylor K. Developing and validating the Communication Function Classification System for individuals with cerebral palsy. Dev Med Child Neurol. 2011 Aug;53(8):704-10. doi: 10.1111/j.1469-8749.2011.03996.x. Epub 2011 Jun 27. PMID 21707596
- [Background] Fox MA, Ayyangar R, Parten R, Haapala HJ, Schilling SG, Kalpakjian CZ. Self-report of pain in young people and adults with spastic cerebral palsy: interrater reliability of the revised Face, Legs, Activity, Cry, and Consolability (r-FLACC) scale ratings. Dev Med Child Neurol. 2019 Jan;61(1):69-74. doi: 10.1111/dmcn.13980. Epub 2018 Jul 27. PMID 30051908
- [Background] Caravau H, Rosa AF, Rocha NP, Silva AG. Pain assessment in cerebral palsy: a systematic review of measurement properties and evaluation using the COSMIN checklist. Disabil Rehabil. 2022 Mar;44(6):910-920. doi: 10.1080/09638288.2020.1783000. Epub 2020 Jul 3. PMID 32619368
- [Background] Boldingh EJ, Jacobs-van der Bruggen MA, Lankhorst GJ, Bouter LM. Assessing pain in patients with severe cerebral palsy: development, reliability, and validity of a pain assessment instrument for cerebral palsy. Arch Phys Med Rehabil. 2004 May;85(5):758-66. doi: 10.1016/j.apmr.2003.06.029. PMID 15129400
- [Background] Letzkus L, Fehlings D, Ayala L, Byrne R, Gehred A, Maitre NL, Noritz G, Rosenberg NS, Tanner K, Vargus-Adams J, Winter S, Lewandowski DJ, Novak I. A Systematic Review of Assessments and Interventions for Chronic Pain in Young Children With or at High Risk for Cerebral Palsy. J Child Neurol. 2021 Aug;36(9):697-710. doi: 10.1177/0883073821996916. Epub 2021 Mar 9. PMID 33719661
- [Background] Jozwiak M, Harasymczuk P, Koch A, Kotwicki T. Incidence and risk factors of hip joint pain in children with severe cerebral palsy. Disabil Rehabil. 2011;33(15-16):1367-72. doi: 10.3109/09638288.2010.532281. Epub 2010 Nov 20. PMID 21091045
- [Background] Faccioli S, Sassi S, Ferrari A, Corradini E, Toni F, Kaleci S, Lombardi F, Picelli A, Benedetti MG. Prevalence and determinants of hip pain in non-ambulatory cerebral palsy children: a retrospective cohort study. Eur J Phys Rehabil Med. 2023 Feb;59(1):32-41. doi: 10.23736/S1973-9087.22.07725-5. Epub 2022 Dec 12. PMID 36507793
- [Background] Jayanath S, Ong LC, Marret MJ, Fauzi AA. Parent-reported pain in non-verbal children and adolescents with cerebral palsy. Dev Med Child Neurol. 2016 Apr;58(4):395-401. doi: 10.1111/dmcn.12943. Epub 2015 Oct 28. PMID 26510627
- [Background] Kingsnorth S, Orava T, Provvidenza C, Adler E, Ami N, Gresley-Jones T, Mankad D, Slonim N, Fay L, Joachimides N, Hoffman A, Hung R, Fehlings D. Chronic Pain Assessment Tools for Cerebral Palsy: A Systematic Review. Pediatrics. 2015 Oct;136(4):e947-60. doi: 10.1542/peds.2015-0273. PMID 26416940
- [Background] Penner M, Xie WY, Binepal N, Switzer L, Fehlings D. Characteristics of pain in children and youth with cerebral palsy. Pediatrics. 2013 Aug;132(2):e407-13. doi: 10.1542/peds.2013-0224. Epub 2013 Jul 15. PMID 23858420
- [Background] Ostojic K, Paget S, Kyriagis M, Morrow A. Acute and Chronic Pain in Children and Adolescents With Cerebral Palsy: Prevalence, Interference, and Management. Arch Phys Med Rehabil. 2020 Feb;101(2):213-219. doi: 10.1016/j.apmr.2019.08.475. Epub 2019 Sep 12. PMID 31521713